CLINICAL TRIAL: NCT04722406
Title: Tumor Growth Rate (TGR) as an Early Predictor of Clinical Outcomes in Advanced Non-small Cell Lung Cancer Treated With PD-1 Axis Inhibitors.
Brief Title: Tumor Growth Rate (TGR) Predicts Clinical Outcomes for Advanced Non-small Cell Lung Cancer Undergoing Immunotherapy.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Shaodong Hong, Deputy Chief Physician, MD, Sun Yat-sen University
Other Study IDs: SHong
Record Dates: First submitted 2021-01-18; First posted 2021-01-25 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Tumor Growth Rate; NSCLC; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low TGR group: Patients with low level of TGR determined by X-tile program
  Interventions: Other: This item is not applicable to our observational study.
- High TGR group: Patients with high level of TGR determined by X-tile program
  Interventions: Other: This item is not applicable to our observational study.

INTERVENTIONS:
Other: This item is not applicable to our observational study. — This item is not applicable to our observational study.

SUMMARY:
We hypothesized that TGR could serve as an early predictor of outcomes for aNSCLC patients undergoing immune checkpoint inhibitors (ICIs). A retrospective analysis was conducted to investigate the association of TGR with response and long-term survival of aNSCLC patients undergoing ICI therapy.

DETAILED DESCRIPTION:
Tumor growth rate (TGR) signifies percentage change in tumor size per month (%/m). Electronic medical records were retrospectively reviewed for all histologically confirmed aNSCLC patients undergoing anti-PD-1/PD-L1 therapy at Sun Yat-Sen University Cancer Center (SYSUCC) between August 2016 and June 2018.

All response and outcome evaluation were determined as per RECIST 1.1 by two senior radiologists blinded to patients'information. Discrepancy was solved by consensus.

X-tile software was used to determine cut-off values that maximumly differentiate overall survival (OS). Log-rank tests and Cox regression models were performed for survival analysis. The predictive value of TGR for clinical outcomes in ICI-treated aNSCLC patients was validated in two external cohorts, recruited form Guangdong Province Traditional Chinese Medical Hospital and Shanghai Chest Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed aNSCLC patients
* Having received anti-PD-1/PD-L1 therapy
* Must have two consecutive computed tomography (CT) scans upon early treatment (from baseline to the first imaging evaluation)

Exclusion Criteria:

* Lacking available computed tomography (CT) evaluation at any of two time points-baseline and the first evaluation
* Without measurable lesions at baseline CT scan
* Having received local anticancer therapy during ICI treatment, for example, radiotherapy and radiofrequency ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All histologically confirmed aNSCLC patients undergoing anti-PD-1/PD-L1 therapy (N = 172) at Sun Yat-Sen University Cancer Center (SYSUCC) between August 2016 and June 2018.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival of patients undergoing ICI monotherapy | From date of ICI treatment initiation until the date of death from any causes, assessed up to 100 months.
  Overall survival (OS) was defined as the time from immunotherapy initiation to death from any causes.

SECONDARY OUTCOMES:
Progression-free survival of patients undergoing ICI monotherapy. | From date of ICI treatment initiation until the date of first documented progression or date of death from any causes, whichever came first, assessed up to 100 months.
  Progression-free survival was calculated from ICI initiation to radiologically-defined progression or death from any causes.

CONTACTS AND LOCATIONS:
Overall Officials: Shaodong Hong, MD, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Shaihai Chest Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
Data including demographic characteristics, clinical information, radiological and follow-up information will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: The IPD and any additional supporting information will become available 3 months after publication.
Access Criteria: data can be obtained from the principal investigator by e-mail upon reasonable request.

REFERENCES:
- [Background] Antonia SJ, Borghaei H, Ramalingam SS, Horn L, De Castro Carpeno J, Pluzanski A, Burgio MA, Garassino M, Chow LQM, Gettinger S, Crino L, Planchard D, Butts C, Drilon A, Wojcik-Tomaszewska J, Otterson GA, Agrawal S, Li A, Penrod JR, Brahmer J. Four-year survival with nivolumab in patients with previously treated advanced non-small-cell lung cancer: a pooled analysis. Lancet Oncol. 2019 Oct;20(10):1395-1408. doi: 10.1016/S1470-2045(19)30407-3. Epub 2019 Aug 14. PMID 31422028
- [Background] Xia L, Liu Y, Wang Y. PD-1/PD-L1 Blockade Therapy in Advanced Non-Small-Cell Lung Cancer: Current Status and Future Directions. Oncologist. 2019 Feb;24(Suppl 1):S31-S41. doi: 10.1634/theoncologist.2019-IO-S1-s05. PMID 30819829
- [Background] Mok TSK, Wu YL, Kudaba I, Kowalski DM, Cho BC, Turna HZ, Castro G Jr, Srimuninnimit V, Laktionov KK, Bondarenko I, Kubota K, Lubiniecki GM, Zhang J, Kush D, Lopes G; KEYNOTE-042 Investigators. Pembrolizumab versus chemotherapy for previously untreated, PD-L1-expressing, locally advanced or metastatic non-small-cell lung cancer (KEYNOTE-042): a randomised, open-label, controlled, phase 3 trial. Lancet. 2019 May 4;393(10183):1819-1830. doi: 10.1016/S0140-6736(18)32409-7. Epub 2019 Apr 4. PMID 30955977
- [Background] Gettinger S, Horn L, Jackman D, Spigel D, Antonia S, Hellmann M, Powderly J, Heist R, Sequist LV, Smith DC, Leming P, Geese WJ, Yoon D, Li A, Brahmer J. Five-Year Follow-Up of Nivolumab in Previously Treated Advanced Non-Small-Cell Lung Cancer: Results From the CA209-003 Study. J Clin Oncol. 2018 Jun 10;36(17):1675-1684. doi: 10.1200/JCO.2017.77.0412. Epub 2018 Mar 23. PMID 29570421
- [Background] Ferte C, Fernandez M, Hollebecque A, Koscielny S, Levy A, Massard C, Balheda R, Bot B, Gomez-Roca C, Dromain C, Ammari S, Soria JC. Tumor growth rate is an early indicator of antitumor drug activity in phase I clinical trials. Clin Cancer Res. 2014 Jan 1;20(1):246-52. doi: 10.1158/1078-0432.CCR-13-2098. Epub 2013 Nov 15. PMID 24240109
- [Background] Lamarca A, Crona J, Ronot M, Opalinska M, Lopez Lopez C, Pezzutti D, Najran P, Carvhalo L, Franca Bezerra RO, Borg P, Vietti Violi N, Vidal Trueba H, de Mestier L, Schaefer N, Sundin A, Costa F, Pavel M, Dromain C; Knowledge Network. Value of Tumor Growth Rate (TGR) as an Early Biomarker Predictor of Patients' Outcome in Neuroendocrine Tumors (NET)-The GREPONET Study. Oncologist. 2019 Nov;24(11):e1082-e1090. doi: 10.1634/theoncologist.2018-0672. Epub 2019 Mar 25. PMID 30910869
- [Background] Stein WD, Wilkerson J, Kim ST, Huang X, Motzer RJ, Fojo AT, Bates SE. Analyzing the pivotal trial that compared sunitinib and IFN-alpha in renal cell carcinoma, using a method that assesses tumor regression and growth. Clin Cancer Res. 2012 Apr 15;18(8):2374-81. doi: 10.1158/1078-0432.CCR-11-2275. Epub 2012 Feb 17. PMID 22344231
- [Background] Gomez-Roca C, Koscielny S, Ribrag V, Dromain C, Marzouk I, Bidault F, Bahleda R, Ferte C, Massard C, Soria JC. Tumour growth rates and RECIST criteria in early drug development. Eur J Cancer. 2011 Nov;47(17):2512-6. doi: 10.1016/j.ejca.2011.06.012. Epub 2011 Jul 15. PMID 21763126
- [Background] Camp RL, Dolled-Filhart M, Rimm DL. X-tile: a new bio-informatics tool for biomarker assessment and outcome-based cut-point optimization. Clin Cancer Res. 2004 Nov 1;10(21):7252-9. doi: 10.1158/1078-0432.CCR-04-0713. PMID 15534099
- [Derived] He LN, Fu S, Ma H, Chen C, Zhang X, Li H, Du W, Chen T, Jiang Y, Wang Y, Wang Y, Zhou Y, Lin Z, Yang Y, Huang Y, Zhao H, Fang W, Zhang H, Zhang L, Hong S. Early on-treatment tumor growth rate (EOT-TGR) determines treatment outcomes of advanced non-small-cell lung cancer patients treated with programmed cell death protein 1 axis inhibitor. ESMO Open. 2022 Dec;7(6):100630. doi: 10.1016/j.esmoop.2022.100630. Epub 2022 Nov 25. PMID 36442353